CLINICAL TRIAL: NCT01031043
Title: Topical Bethanechol for Improvement of Esophageal Dysmotility: A Pilot Study
Brief Title: Topical Bethanechol for Improvement of Esophageal Dysmotility
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Gregory Postma, Professor, Augusta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-03-244
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2015-01-29 (Estimated); Last update posted 2015-01-29 (Estimated); Status verified 2015-01

CONDITIONS: Esophageal Dysmotility
Keywords: IEM
MeSH Terms: conditions — Esophageal Motility Disorders | interventions — Bethanechol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Topical Bethanechol (Experimental): patients will be given either 5 mg (first phase) or 10 mg (second phase) of bethanechol in 1 ml of solution containing an absorption enhancer. Administration will be performed by throat spray device
  Interventions: Drug: Bethanechol

INTERVENTIONS:
Drug: Bethanechol — Taking part in this research study is voluntary. Patient may choose not to take part in this research study or may withdraw consent at any time. Their choice will not at any time affect the commitment of the health care providers to administer care. If the patient decides not to participate or withdraw from the study there will be no penalty or loss of benefits to which they are otherwise entitled.
  Other Names: Urecholine

SUMMARY:
The purpose of this research project is to determine the effect of a drug called bethanechol on swallowing function in patients with Ineffective Esophageal Motility (IEM). This drug is FDA approved for use in treating other conditions, but not for the treatment of IEM. There is currently no approved therapy for the treatment of IEM. This information is important for the possible development of new ways of treating patients with IEM and for the effectiveness of topically applied Bethanechol on patients with IEM.

DETAILED DESCRIPTION:
This is a pilot study, and as such is not necessarily expected to achieve statistical significance. A control group will not be used, again owing to the pilot nature of the study. Previous studies have demonstrated the safety of oral bethanechol. It has shown some efficacy in the treatment of gastroesophageal reflux in both adults and children1-8, and there is extensive preclinical data suggesting a beneficial effect for patients with IEM9-14. A single study15 of oral bethanechol in patients with IEM demonstrated a significant improvement in distal esophageal muscle contraction and bolus transit. This study, however measured esophageal function using an inferior method of manometry. The proposed study uses high-resolution manometry to measure the effects of oral bethanechol in patients with IEM, and will yield improved understanding of changes in esophageal function in real-time. The study intervention (oral bethanechol) will be a single-dose event (applied in two encounters), not an ongoing treatment intervention.

We will evaluate the effect of topically applied bethanechol on esophageal motility in a cohort (n=20) of patients with IEM. Presence of IEM will be defined using current criteria: esophageal contraction amplitude <30 mmHg either 5 or 10 cm above the lower esophageal sphincter, in 50% or more of saline swallows15, 16. We will perform high-resolution manometry (HRM) to establish a baseline in these patients. HRM is part of the cutting-edge technology available at the Medical College of Georgia Center for Voice and Swallowing Disorders (CVSD, part of the Department of Otolaryngology), and is used in the clinical evaluation of patients with dysphagia on a routine basis. Many patients with IEM referred to the CVSD will undergo high-resolution manometry during the course of their evaluation and treatment, regardless of inclusion in this study. The test consists of placement of a manometry catheter through the nasal cavity into the esophagus, much as a naso-gastric tube would be placed. After confirming proper placement of the catheter by manometry, the patient is asked to perform 10 swallows of a teaspoon (5ml) of water. The muscle contractions of the esophagus, including the upper and lower esophageal sphincters, are then recorded in real-time along the entire length of the catheter for the duration of the swallow. This allows measurement and analysis of not only isolated contraction events, but also the entire swallow as it propagates down the esophagus.

Following establishment of baseline esophageal function, patients will be given either 5 mg (first phase) or 10 mg (second phase) of bethanechol in 1 ml of solution containing an absorption enhancer. Administration will be performed by throat spray device. The composition of the delivery solution is proprietary. Since bethanechol is a quaternary amine known to have less than 1 % topical absorbance, an absorption enhancer is necessary to aid in this process. The choice of an appropriate FDA approved absorption enhancer is what makes this preparation unique. The preparation also contains thickening agents that allow it to remain where sprayed to enhance absorption.

After waiting 10 minutes, patients will then undergo a post-treatment HRM to establish treatment effect. The manometry catheter will be left in place during the entire encounter, thus requiring only the single placement of the catheter per sessions. Two sessions will be required to establish dose escalation effect.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient treated at the Medical College of Georgia, with severe IEM as defined using current criteria: esophageal contraction amplitude <30 mmHg either 5 or 10 cm above the lower esophageal sphincter, in 50% or more of saline swallows.

Exclusion Criteria:

* Patients with severe comorbidities (including uncontrolled hypertension, severe coronary artery disease, and uncontrolled diabetes) will be specifically excluded from the study.
* Additionally, the use of bethanechol (as well as all other muscarinic receptor agonists) is contraindicated in patients with asthma, coronary insufficiency, peptic ulcers, Parkinson's disease, seizure disorder, recent gastrointestinal surgery, and hyperthyroidism. As such any patient with these disorders will be specifically excluded from this study.
* Women of childbearing age will also be specifically excluded (Bethanechol is listed as a pregnancy class C drug).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory N Postma, MD, Principal Investigator — Augusta University
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult volunteers with a diagnosis of Esophageal Dysmotility were recruited from the senior author's clinical practice.
Period: Overall Study
Arm/Group | Topical Bethanechol
Started | 5
Completed | 4
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Topical Bethanechol
Number analyzed (Participants) | 5
Age, Continuous [Median (Standard Deviation); unit: years] | 48 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Distal Contractile Integral
Description: The index of contractile strength of the esophageal smooth muscle. The range of the index being 0 mmHg *s*cm to >10,000 mmHg *s*cm where 0 represents no contractile strength. The index reflects the magnitude of distal esophageal contraction, taking into consideration the length, strength, and duration of the contraction.
Time Frame: Encounter 1 (day 1) and Encounter 2 (Month 14)
Population: All subjects enrolled in the study
Measure: Mean (Standard Deviation); unit: mmHg*s*cm
Arm/Group | Topical Bethanechol
Number analyzed (Participants) | 5
mmHg*s*cm
  Baseline Measure | 178.3 (83.1)
  5 mg dose of Bethanechol | 272.3 (216.9)
  10 mg dose of Bethanechol | 261.8 (293.5)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Topical Bethanechol
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No